CLINICAL TRIAL: NCT06292845
Title: Ex Vivo Tumor Visualization and Resection Margin Assessment Using Topically Applied Fluorescent Imaging Agents
Acronym: SprayDye
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Stijn Keereweer, Dr., Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 11272
Record Dates: First submitted 2023-11-20; First posted 2024-03-05 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Solid Tumor, Adult
Keywords: Fluorescence imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Topical application of a fluorescent imaging agent (Experimental): In this arm the investigators use the freshly resected human solid tumor specimens to assess the performance of topically applied fluorescent imaging agents for the detection of tumor tissue and close / tumor-positive resection margins ex vivo.
  Interventions: Drug: Topical application of a fluorescent imaging agent

INTERVENTIONS:
Drug: Topical application of a fluorescent imaging agent — The fluorescent imaging agent will be topically applied only onto the resection planes of the freshly resected tumor specimen.
  During incubation and after each washing steps, visible light and fluorescent overlay images will be acquired using a fluorescence sensitive camera system.
  Other Names: fluorescent imaging agent

SUMMARY:
This is a proof-of-principle study, that uses freshly resected human solid tumor specimens to assess the performance of topically applied fluorescent imaging agents for the detection of tumor tissue and close / tumor-positive resection margins ex vivo. Surgery will be performed in conformity with hospital protocol. The study will not interfere with the standard clinical care.

DETAILED DESCRIPTION:
Surgical excision remains an integral part of curative-intent treatment for most solid tumors. The goal of surgical resection is to completely remove all tumor tissue. A tumor-positive or inadequate surgical resection margin, defined as cancer cells at or near (depending on tumor type) the edge of the resection specimen, has major prognostic implications and often necessitates additional treatments. These additional treatments are in turn associated with increased morbidity, complication risks, and healthcare costs.

To achieve a complete resection of the tumor, surgeons rely on visual inspection and palpation, sometimes assisted by localization or pathology techniques such as implanted (radioactive/magnetic) seeds and frozen section analysis. However, inadequate resection margin rates in solid tumors remain high, indicating current methods for intraoperative margin assessment are insufficient. They lack real-time feedback on the margin status of large tissue surface areas to guide additional resection.

A technique that could meet these requirements is tumor-targeted fluorescence imaging (FI). It combines the administration of a fluorescence imaging agent with the use of fluorescence light. This technique allows for real-time optical feedback by selectively highlighting tumor tissue that expresses certain molecular targets that bind the imaging agent or has certain characteristics that activate it.

Presently, the vast majority of fluorescence imaging agents under investigation for intraoperative tumor visualization and resection margin assessment have to be administered intravenously, hours or days prior to surgery. Very recently, new imaging agents have been designed that can be topically administered. Topically applied imaging agents allow for specimen-based (ex vivo) resection-margin assessment using FI, without the necessity to administer the probe to the patient. This approach offers several advantages: (I) ex vivo topical application on the resected specimen eliminates all toxicity risks, as the patient is not exposed to the imaging agent; (II) it is much more cost-effective. First of all, a lower imaging agent dose can be used because there is no systemic volume of distribution, and the probe is not metabolized and excreted. Secondly, toxicity testing and in-patient clinical trials are not required to use the ex vivo topical approach in clinical practice, which greatly reduces implementation time and costs; (III) the ex vivo topical approach is easier to implement in the current surgical workflow, and does not require the patient logistics needed for systemic administration.

In this proof-of-principle study, the investigators will investigate if topically applied fluorescent imaging agents can be used to visualize tumor tissue and detect inadequate resection margins ex vivo on freshly resected solid human tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a biopsy-proven solid tumor, scheduled for surgery at the Erasmus Medical Center.
2. Signed and dated informed consent obtained before any study-related procedure is performed.

Exclusion Criteria:

1. Terminated surgical procedure.
2. No fresh specimen available.
3. Participation in a clinical trial for which the patient receives another fluorophore perioperatively.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-01-16 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Tumor-to-background ratio (TBR) of the fluorescence signal on the resection specimen surface and on 3-5 mm thick tissue slices. | through study completion, up to 3 years
  TBR was calculated by drawing a region of interest (ROI) spanning the tumor, and another in adjacent (muscle) tissue using the imaging system's integrated software

SECONDARY OUTCOMES:
Imaging agent fluorescence signal intensity on close / tumor-positive resection planes compared with (wide) tumor-negative resection planes, as confirmed by histopathology | through study completion, up to 3 years
  Signal intensity was determined from a region of interest (ROI) drawn in close / tumor-positive resection planes as well as (wide) tumor-negative resection planes, and comparing them using the imaging system's integrated software.
Difference in tumor-to-background ratio (TBR) between different imaging time windows | through study completion, up to 3 years
  TBR was calculated for different imaging time windows, and compared.
The concordance between the presence of tumor cells and fluorescence signal | through study completion, up to 3 years
  Overlaying fluorescence images with corresponding H&E slides
Depth of the fluorescence signal on 4-μm tissue slides | through study completion, up to 3 years
  Penetration depth of topically applied fluorescent imaging agents was determined from fluorescence images

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus University Medical Center, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes